CLINICAL TRIAL: NCT06205589
Title: A Phase 2a/2b Study Evaluating Safety, Immunogenicity, and Therapeutic Efficacy of ID93 + GLA-SE Vaccination in Participants With Rifampicin-Susceptible Pulmonary TB
Brief Title: Therapeutic ID93 + GLA-SE Vaccination in Participants With Rifampicin-Susceptible Pulmonary TB
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5397; UM1AI068636 (NIH)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Group 1/Phase 2a: ID93+GLA-SE 4 months and 6 months after start of TB treatment (Active Comparator): Participants will be enrolled at approximately 4 months after the start of TB treatment, entering the study directly into Step 2, and will be randomized to receive ID93 + GLA-SE immediately. They have no Step 1 observation period from the start of SOC TB treatment to randomization.
  Interventions: Biological: ID93 + GLA-SE vaccine
- Group 2/Phase 2a: ID93+GLA-SE 3 months and 5 months after start of TB treatment (Active Comparator): Participants will be enrolled at approximately 3 months after the start of TB treatment, entering the study directly into Step 2, and will be randomized to receive ID93 + GLA-SE or placebo immediately. They have no Step 1 observation period from the start of SOC TB treatment to randomization.
  Interventions: Biological: ID93 + GLA-SE vaccine
- Group 3/Phase 2a: ID93+GLA-SE 2 months and 4 months after start of TB treatment (Active Comparator): Participants will enter the study within approximately 7 days after starting TB treatment in Step 1, which is an observation period between the start of SOC TB treatment until entering Step 2. In Step 2 they will be randomized to ID93 + GLA-SE at 2 months after study entry/start of TB treatment.
  Interventions: Biological: ID93 + GLA-SE vaccine
- Group 4/Phase 2a: ID93+GLA-SE 1 month and 3 months after start of TB treatment (Active Comparator): Participants will enter the study within approximately 7 days after starting TB treatment in Step 1, which is an observation period between the start of SOC TB treatment until entering Step 2. In Step 2 they will be randomized to ID93 + GLA-SE 1 month after study entry/start of TB treatment.
  Interventions: Biological: ID93 + GLA-SE vaccine
- Group 5/Phase 2b: ID93+GLA-SE schedule based on Group 3 and 4 safety and immunogenicity data (Active Comparator): Participants will enter the study within approximately 7 days after starting TB treatment in Step 1, which is an observation period between the start of SOC TB treatment until entering Step 2. The vaccination schedule will be selected from either the Group 3 or Group 4 schedule, following a review of the safety and immunogenicity data after the last participant in Group 4 receives the second vaccination. If both the safety and immunogenicity criteria are met, the Group 4 schedule will be selected and Group 5 will include Group 4 participants. If Group 4 fails to meet both the safety and immunogenicity criteria, the Group 3 vaccination schedule will be selected and Group 5 will include Group 3 participants. If safety and immunogenicity criteria are not met in either Group 3 or 4, then enrollment to Group 5 will not proceed and the phase 2b component of the study will not be undertaken.
  Interventions: Biological: ID93 + GLA-SE vaccine
- Group 1/Phase 2a: Placebo vaccine 4 months and 6 months after start of TB treatment (Placebo Comparator): Participants will be enrolled at approximately 4 months after the start of TB treatment, entering the study directly into Step 2, and will be randomized to receive placebo immediately. They have no Step 1 observation period from the start of SOC TB treatment to randomization.
  Interventions: Biological: Placebo vaccine
- Group 2/Phase 2a: Placebo vaccine 3 months and 5 months after start of TB treatment (Placebo Comparator): Participants will be enrolled at approximately 3 months after the start of TB treatment, entering the study directly into Step 2, and will be randomized to receive placebo immediately. They have no Step 1 observation period from the start of SOC TB treatment to randomization.
  Interventions: Biological: Placebo vaccine
- Group 3/Phase 2a: Placebo vaccine 2 months and 4 months after start of TB treatment (Placebo Comparator): Participants will enter the study within approximately 7 days after starting TB treatment in Step 1, which is an observation period between the start of SOC TB treatment until entering Step 2. In Step 2 they will be randomized to placebo at 2 months after study entry/start of TB treatment.
  Interventions: Biological: Placebo vaccine
- Group 4/Phase 2a: Placebo vaccine 1 month and 3 months after start of TB treatment (Placebo Comparator): Participants will enter the study within approximately 7 days after starting TB treatment in Step 1, which is an observation period between the start of SOC TB treatment until entering Step 2. In Step 2 they will be randomized to ID93 + GLA-SE or placebo 1 month after study entry/start of TB treatment.
  Interventions: Biological: Placebo vaccine
- Group 5/Phase 2b: Placebo vaccine schedule based on Group 3 and 4 safety and immunogenicity data (Placebo Comparator): Participants will enter the study within approximately 7 days after starting TB treatment in Step 1, which is an observation period between the start of SOC TB treatment until entering Step 2. The vaccination schedule will be selected from either the Group 3 or Group 4 schedule, following a review of the safety and immunogenicity data after the last participant in Group 4 receives the second vaccination. If both the safety and immunogenicity criteria are met, the Group 4 schedule will be selected and Group 5 will include Group 4 participants. If Group 4 fails to meet both the safety and immunogenicity criteria, the Group 3 vaccination schedule will be selected and Group 5 will include Group 3 participants. If safety and immunogenicity criteria are not met in either Group 3 or 4, then enrollment to Group 5 will not proceed and the phase 2b component of the study will not be undertaken.
  Interventions: Biological: Placebo vaccine

INTERVENTIONS:
Biological: ID93 + GLA-SE vaccine — At Step 2 entry, participants will receive one 0.5 mL injection of ID93 + GLA-SE administered intramuscularly (IM) at the Step 2, Day 0 visit and at the Step 2, Day 60 visit per the dosing schedule within the respective group/arm.
  Arms: Group 1/Phase 2a: ID93+GLA-SE 4 months and 6 months after start of TB treatment; Group 2/Phase 2a: ID93+GLA-SE 3 months and 5 months after start of TB treatment; Group 3/Phase 2a: ID93+GLA-SE 2 months and 4 months after start of TB treatment; Group 4/Phase 2a: ID93+GLA-SE 1 month and 3 months after start of TB treatment; Group 5/Phase 2b: ID93+GLA-SE schedule based on Group 3 and 4 safety and immunogenicity data
Biological: Placebo vaccine — At Step 2 entry, participants will receive one placebo injection (sodium Chloride, 0.9%) administered intramuscularly (IM) at the Step 2, Day 0 visit and at the Step 2, Day 60 visit per the dosing schedule within the respective group/arm.
  Arms: Group 1/Phase 2a: Placebo vaccine 4 months and 6 months after start of TB treatment; Group 2/Phase 2a: Placebo vaccine 3 months and 5 months after start of TB treatment; Group 3/Phase 2a: Placebo vaccine 2 months and 4 months after start of TB treatment; Group 4/Phase 2a: Placebo vaccine 1 month and 3 months after start of TB treatment; Group 5/Phase 2b: Placebo vaccine schedule based on Group 3 and 4 safety and immunogenicity data

SUMMARY:
This study is being done to test an experimental study vaccine compared to a placebo. The experimental study vaccine is called ID93 + GLA-SE. ID93 + GLA-SE has been used in humans in research but has not been approved for use in medical care. This study will be the first to test ID93 + GLA-SE in people living with HIV (PLWH). The injections during the study will be given to different groups of participants while they are using standard TB treatment. One of the research questions is to understand the differences in immune system responses depending on the timing of giving the injections after people begin taking standard TB treatment. Researchers also want to continue to look at whether the study vaccine is safe when tested in a larger group of people, and if getting the study vaccine in addition to standard TB treatment can help to lower the number of poor TB outcomes that people might have.

ELIGIBILITY:
Inclusion Criteria Groups 1-5:

* Bacteriologically confirmed rifampicin-susceptible pulmonary TB using phenotypic drug susceptibility testing or a World Health Organization (WHO) approved molecular test.
* Documentation of HIV status as positive or negative by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit.
* For individuals with HIV, on locally approved HIV ART for at least 90 days prior to entry.
* For individuals with HIV, CD4+ cell count ≥250 cells/mm3 obtained within 90 days prior to entry at any network-approved non-US laboratory that is DAIDS IQA certified.
* For individuals with HIV, HIV-1 RNA below the limit of detection obtained within 90 days prior to entry by any network-approved laboratory outside the US that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance programs.
* Laboratory values within the indicated ranges, obtained within 14 days prior to entry by any network-approved laboratory outside the US that operates in accordance with GCLP and participates in appropriate external quality assurance programs.

  * Absolute neutrophil count (ANC) ≥800 cells/mm3
  * Hemoglobin ≥8.5 g/dL for candidates assigned female sex at birth and >9.0 g/dL for candidates assigned male sex at birth
  * Platelet count ≥100,000/mm3
  * Serum creatinine ≤1.5 X upper limit of normal (ULN)
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase, ≤2.5 X ULN
  * Total bilirubin ≤2 X ULN
* For candidates who are able to become pregnant, negative serum or urine pregnancy test at or within 7 days prior to entry by any network-approved laboratory or clinic outside the US that operates in accordance with GCLP and participates in appropriate external quality assurance programs.
* Candidates who are able to become pregnant must agree to use an adequate method of contraception (barrier methods or non-hormonal intrauterine device) or abstain from sexual activity that could lead to pregnancy from at least 21 days prior to the first scheduled vaccination through 90 days after last dose.
* Candidates assigned female sex at birth (AFAB) must agree to not seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination, or in vitro fertilization, from at least 21 days prior to the first scheduled vaccination through 90 days after last dose.
* For candidates who are not of child-bearing potential, acceptable documentation (written documentation or oral communication from a clinician or clinician's staff documented in source documents: physician report/letter, operative report or other source documentation in the candidate record, discharge summary, laboratory report, etc.) of hysterectomy and bilateral oophorectomy, tubal ligation, tubal micro-inserts, vasectomy, or menopause.
* Ability and willingness of candidate to provide informed consent.

Inclusion Criteria Groups 1 and 2 [Step 2]:

* Documented duration of local SOC TB treatment prior to entry into Step 2 (study entry) for i. Group 1 of between 113 and 127 days (i.e., approximately 4 months of TB treatment) ii. Group 2 of between 83 and 97 days (i.e., approximately 3 months of TB treatment)

Inclusion Criteria, Groups 3, 4, and 5 [Step 1]:

* Initiation of local SOC TB treatment within 7 days prior to entry into Step 1 (Study entry).

Exclusion Criteria Groups 1-5:

* Documented M.tb resistance to isoniazid.
* Breastfeeding.
* Any previous episode of TB treatment.
* TB treatment with a local non-standard first-line TB treatment regimen at time of enrollment.
* Receipt of any investigational drug or any investigational non-TB vaccine since start of TB treatment.
* Any prior receipt of any investigational TB vaccine.
* Known allergy or any hypersensitivity to any components of study product or their formulation or any vaccination.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* History of moderate to serious autoimmune disease requiring immunosuppressive therapy.
* Receipt of immunosuppressive medications (except as noted below) from start of TB treatment.

  * Corticosteroid nasal spray
  * Inhaled corticosteroids
  * Topical corticosteroids for mild, uncomplicated dermatologic condition
  * A single course of oral/parenteral prednisone or equivalent at doses <60 mg/day and for <11 days with completion at least 30 days prior to entry.
* Receipt of Emergency Use Authorization (EUA)/Emergency Use Listing (EUL) or licensed live attenuated vaccines (e.g., measles, mumps, and rubella [MMR], oral polio vaccine [OPV], varicella, yellow fever, live attenuated influenza vaccine, live attenuated COVID-19 vaccine) within 30 days prior to entry.
* Receipt of any EUA/EUL or licensed vaccines that are not live attenuated vaccines (e.g., tetanus, pneumococcal, Hepatitis A or B, not live attenuated COVID-19 vaccine) within 14 days prior to entry.
* Receipt of immunoglobulin or blood-derived products within 90 days prior to entry.
* History of angioedema, or anaphylaxis, except as noted.
* History of generalized urticaria within past 5 years.
* Malignancy, except as noted.
* Daily (current) use of a short-acting rescue inhaler (e.g., a beta 2 agonist).
* Within the previous year, exacerbation of asthma symptoms requiring emergency care, urgent care, hospitalization, or intubation.
* Uncontrolled diabetes mellitus type 1 or type 2, defined as Hemoglobin A1c (HbA1C) >7%.
* Bleeding disorder (e.g., factor deficiency, coagulopathy, platelet disorder requiring special precautions).
* Seizure disorder, including either of the following within the previous 3 years:

  * Seizure(s)
  * Use of medications to prevent or treat seizure(s)
* Acute or serious illness, including COVID-19, requiring systemic treatment and/or hospitalization from start of TB treatment, other than for pulmonary TB.
* Documentation of clinically significant (as judged by the site investigator) active infections (including HIV-related opportunistic infections) other than TB and HIV requiring treatment within 30 days prior to entry.
* Evidence of clinically significant disease (as judged by the site investigator) or any other abnormalities (other than the indication being studied) that would interfere with study product, procedures, or interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
* Suspected or documented TB involving the central nervous system, renal TB or TB pericarditis, or current extrapulmonary TB involving other organ systems that might interfere with study product or procedures, as judged by the site investigator.
* Contraindication to intramuscular injection in both deltoids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-10-13 (Estimated)

PRIMARY OUTCOMES:
Safety (Phase 2a and Phase 2b): Vaccine-related serious adverse event (SAE) | From Step 2, Day 0 through to 420, 450, 480 or 510 days (approximately 18 months after start of SOC treatment)
  Vaccine-related serious adverse event (SAE) at any time after first dose of ID93 + GLA-SE. The relationship to study product will be determined by the site investigator and assessed as "related" or "unrelated". Only SAEs reported as "related" will be included in this outcome measure.
Safety (Phase 2a and Phase 2b): Grade ≥3 vaccine-related unsolicited adverse event (AE) | Within 28 days from Step 2, Day 0 or Step 2, Day 60
  Grade ≥3 vaccine-related unsolicited adverse event (AE) within 28 days after either dose of study product. An unsolicited AE is defined as an AE other than a local or systemic reactogenicity AE. The relationship to study product will be determined by the site investigator and assessed as "related" or "unrelated." Only unsolicited AEs reported as "related" will be included in this outcome measure.
Safety (Phase 2a and Phase 2b): Grade ≥3 local or systemic reactogenicity AE | Within 7 days from Step 2, Day 0 or Step 2, Day 60
  o Systemic symptoms include increased body temperature, malaise and/or fatigue, myalgia, headache, chills, arthralgia, nausea, and vomiting. Local symptoms include pain and/or tenderness proximal to the injection site.
Cellular immunogenicity (Phase 2a and Phase 2b): ID93-specific CD4+ T cell response relative to the negative control stimulation | Step 2, Day 75
  ID93-specific CD4+ T cell response relative to the negative control stimulation (ICS response criteria: MIMOSA method) at 2 weeks post second dose of study product. CD4+ T cell response measured by ICS with magnitude indicated by cells expressing 2 of IFNγ/IL2/TNFα/CD154. MIMOSA detects responses compared to the negative control. This will be evaluated as a binary outcome (i.e., response or no response).
Cellular immunogenicity (Phase 2a and Phase 2b): ID93-specific CD4+ T cell response relative to the negative control stimulation and relative to the pre-vaccine response | Step 2, Day 75
  ID93-specific CD4+ T cell response relative to the negative control stimulation and relative to the pre-vaccine response (ICS response criteria: MIMOSA2 method) at 2 weeks post second dose of study product. CD4+ T cell response measured by ICS with magnitude indicated by cells expressing 2 of IFNγ/IL2/TNFα/CD154. MIMOSA2 detects responses compared to the negative control stimulation and the pre-vaccine response. This will be evaluated as a binary outcome (i.e., response or no response).
Cellular immunogenicity (Phase 2a and Phase 2b): ID93-specific CD4+ T cell response magnitude relative to the negative control stimulation | Step 2, Day 75
  ID93-specific CD4+ T cell response magnitude relative to the negative control stimulation at 2 weeks post second dose of study product. CD4+ T cell response measured by ICS with magnitude indicated by cells expressing 2 of IFNγ/IL2/TNFα/CD154. This will be evaluated as a continuous outcome.
Efficacy (Phase 2b): Bacteriologically confirmed TB-related unfavorable outcome (treatment failure, TB recurrence, or death due to TB) | Step 2, Day 0 to 420, 450, 480 or 510 days (approximately 18 months after start of SOC treatment)
  Bacteriologically confirmed TB-related unfavorable outcome (treatment failure, TB recurrence, or death due to TB) after receiving the first dose of study product (ID93 + GLA-SE or placebo). Bacteriological confirmation will be based on culture results from solid media and liquid media that are positive for M. tuberculosis. Culture results from the study or from outside the study (e.g., the local TB program) are acceptable.

SECONDARY OUTCOMES:
Efficacy (Phase 2a and 2b): Proportion of participants with quantifiable RS ratio | Step 2, Days 60, 90, 120, and 150 in Groups 1, 2, 3 (and 5), and 4 (and 5), respectively (approximately 6 months after start of SOC treatment)
  RS ratio will be evaluated as a binary outcome (quantifiable or not quantifiable)
Cellular immunogenicity (Phase 2a): ID93-specific CD4+ T cell response through 12 months post second dose of vaccination | Step 2, Days 0, 15, 60, 75, 120 (Group 3 only), 150 (Group 4 only), 240, 300 (Group 3 only), 330 (Group 4 only) and 420 (Group 2 will be evaluated at Day 450 rather than 420)
  Measured by ICS and flow cytometry. CD4+ T-cell response magnitude indicated by cells expressing 2 of IFNγ/IL2/TNFα/CD154. This will be evaluated as both a binary outcome (response or no response) and as a continuous outcome.
Humoral immunogenicity (Phase 2a): ID93-specific IgG response rate | Step 2, Days 0, 15, 60, 75, 120 (Group 3 only), 150 (Group 4 only), 240, 300 (Group 3 only), 330 (Group 4 only) and 420 (Group 2 will be evaluated at Day 450 rather than 420)
  BAMA response criteria: MFI* >3 x [MFI* at pre-vaccine] and MFI* >100. This will be evaluated as both a binary outcome (i.e., response or no response) and as a continuous outcome.
Immunogenicity (Phase 2a): Differential leukocyte count and immunophenotype | Step 2, Days 0, 1, 15, and 75
  Evaluated in cryopreserved ex vivo whole blood by flow cytometry in Groups 1-4
Immunogenicity (Phase 2a): Measurement of soluble proinflammatory mediators | Step 2, Days 0, 1, 15, and 75
  Evaluated in serum in Groups 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Churchyard, MBBCh, MMED, FCP, PhD, Study Chair — Aurum Institute; James G Kublin, MD, MPH, Study Chair — Fred Hutchinson Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
  Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at:
  https://actgnetwork.org/submit-a-proposal-2/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.